CLINICAL TRIAL: NCT00634413
Title: A Phase II, Randomised, Double-Blind, Placebo-Controlled Pilot Efficacy Study of ADC4022 on Markers of Pulmonary Inflammation in Subjects With Moderate to Severe COPD
Brief Title: Effect of ADC4022 Co-Administered With Budesonide on Pulmonary Inflammation in Subjects With Moderate to Severe COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmagen Therapeutics (Industry)
Responsible Party: Director of Clinical Development, Argenta Discovery Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADC_4022_CLIN_02P
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Theophylline - ADC4022; Drug: Budesonide
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Budesonide

INTERVENTIONS:
Drug: Theophylline - ADC4022 — Inhaled theophylline (ADC4022) administered twice daily for 28 days
  Other Names: ADC4022
  Arms: 1
Drug: Placebo — Inhaled matching placebo administered twice daily for 28 days
  Arms: 2
Drug: Budesonide — Inhaled budesonide twice daily for 28 days
  Other Names: Pulmicort

SUMMARY:
The purpose of this study is to assess the tolerability and efficacy of inhaled theophylline (ADC4022) on markers of pulmonary inflammation (white blood cells) in induced sputum and in bronchial biopsy samples in subjects with moderate to severe Chronic Obstructive Pulmonary Disease (COPD) when co-administered with budesonide and compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COPD that has been symptomatic for at least 2 years
* The subject has moderate to severe COPD, as defined by the American Thoracic Society and the European Respiratory Society
* The subject can produce an adequate sputum specimen after induction
* The subject has a history of ≥ 10-pack years of cigarette smoking
* The subject has either a ≤15% increase or ≤200 ml increase in FEV1 from pre-dose following a fixed dose of bronchodilator therapy
* The subject is able to provide written, informed consent to participate

Exclusion Criteria:

* The subject has experienced a respiratory tract infection and/or an exacerbation of COPD within 30 days
* The subject uses systemic corticosteroids (oral or parenteral)
* The subject has received long term oxygen therapy within 30 days
* The subject has a previous history or diagnosis of asthma
* The subject has a chest x-ray within the past 12 months which is diagnostic of an active or clinically significant disease other than COPD
* The subject has a history or presence of active tuberculosis, cystic fibrosis, bronchiectasis, lung cancer or sarcoidosis or any other clinically important lung diseases
* The subject has had radiation or chemotherapy within the previous 12 months
* The subject has a history of anaphylaxis associated with medicinal products
* The subject is pregnant, intends to become pregnant, or is breast feeding
* The subject's alcohol intake is excessive.
* The subject participated in another study (for a marketed drug) within 3 months before the start of this study or (for an investigational drug) within 4 months before the start of this study.

Other inclusion/exclusion criteria may also apply

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary inflammation: Cell counts (neutrophils, macrophages, eosinophils and lymphocytes) in induced sputum samples | Baseline and after 4 weeks treatment

SECONDARY OUTCOMES:
Pulmonary inflammation: Cytokine IL-8 concentration in induced sputum | Baseline and after 4 weeks treatment
Pulmonary inflammation: CD8+ and CD68+ from bronchial biopsy | Baseline and after 4 weeks treatment
Tolerability to ADC4022 | Baseline, during 4 weeks treatment and after 1 week of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Neil Barnes, MD PhD, Principal Investigator — London Chest Hospital
Locations (8):
- Poland (5):
  - Silisian Medical University, Katowice-Ligota, Katowice-Ligota
  - Jagiellonian University of Medicine, Krakow, Krakow
  - National Tuberculosis and Lung Diseases Research Institute, Warsaw, Warsaw
  - Warsaw University Medical School, Warsaw, Warsaw
  - Medical University in Lodz, Lodz, Łódź Voivodeship
- United Kingdom (3):
  - Glenfield Hospital, Leicester, Leicestershire
  - The London Chest Hospital, London, London
  - Medicines Evaluation Unit, Manchester, Manchester